CLINICAL TRIAL: NCT03816202
Title: Sundt™ Carotid Shunt Retrospective Post Market Clinical Follow-up Study (PMCF)
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-SCS-001
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Sundt Carotid Shunt: Subject has undergone a endarterectomy procedure with the use of the Sundt Carotid Shunt.
  Interventions: Device: Sundt carotid shunt

INTERVENTIONS:
Device: Sundt carotid shunt — The Integra Sundt™ carotid shunts are indicated for temporary carotid artery bypass during carotid endarterectomy procedures to help protect the cerebral hemispheres from ischemia during the period of carotid artery occlusion.

SUMMARY:
The primary objective of this study is to retrospectively investigate the safety and efficacy of the Integra Sundt™ carotid shunt during endarterectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-80 years old
* Have undergone carotid endarterectomy with any Integra Sundt™ carotid shunt on or before date of study initiation
* Availability of records on post-operative imaging of the carotid artery either by carotid duplex ultrasound or angiogram

Exclusion Criteria:

* Insertion of a carotid shunt at the site of an infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in the study have undergone a carotid endarterectomy procedure with the use of the Sundt™ carotid shunt prior to study initiation.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tummon, Study Director — Integra LifeSciences
Locations (3):
- United States (3):
  - Research Institute of Deaconess Clinic, Newburgh, Indiana
  - Hackensack Meridian Health, Hackensack, New Jersey
  - The Mount Sinai Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sundt Carotid Shunt
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sundt Carotid Shunt
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Injury to the Artery or Cerebral Ischemia Secondary to Shunt Placement and Removal
Description: Number of participants with injury to the artery or cerebral ischemia secondary to shunt placement and removal
Time Frame: up to 60 days post-procedure
Population: number of cases where there is evidence of injury to the artery or cerebral ischemia injury secondary to shunt placement and removal
Measure: Count of Participants; unit: Participants
Arm/Group | Sundt Carotid Shunt
Number analyzed (Participants) | 100
Participants | 3

ADVERSE EVENTS:
Time Frame: Retrospective chart review of AEs that occurred between Surgery (Day 0) and 60 days post-operatively.
Groups:
- Sundt Carotid Shunt: number of cases where there is evidence of injury to the artery or cerebral ischemia injury secondary to shunt placement and removal
Arm/Group | Sundt Carotid Shunt
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 3/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sundt Carotid Shunt (N=100)
Cerebral Ischemia Injury (Nervous system disorders) | 2
Artery injury (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT03816202/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT03816202/SAP_001.pdf